CLINICAL TRIAL: NCT01389258
Title: An Open, Prospective, Multi-center Study to Evaluate OsseoSpeed™ TX Single Implant 3 mm Diameter in the Anterior Maxilla. A 3-years Follow-up Study.
Brief Title: Study on OsseoSpeed™ TX Narrow Implants in the Upper Jaw in a Chinese Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dentsply Sirona Implants and Consumables (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHN-0006
Record Dates: First submitted 2011-07-06; First posted 2011-07-08 (Estimated); Results first posted 2019-10-08 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: Partially Edentulous Jaw
MeSH Terms: conditions — Jaw, Edentulous, Partially

ARMS (1):
- OsseoSpeed™ TX (Experimental): OsseoSpeed™ TX narrow implants (diameter 3 mm) of lengths 11-15 mm
  Interventions: Device: OsseoSpeed™ TX

INTERVENTIONS:
Device: OsseoSpeed™ TX — OsseoSpeed™ TX narrow implants (diameter 3 mm) of lengths 11-15 mm

SUMMARY:
The purpose of this study is to investigate the clinical efficacy of OsseoSpeed™ TX 3mm diameter implant in a Chinese population by evaluation of marginal bone level alteration, implant stability and implant survival in the posterior maxilla up to 3 years after loading. Hypothesis: Early loading of the 3 mm implant is a safe and predictable procedure.

ELIGIBILITY:
Inclusion criteria:

1. Provision of informed consent
2. Aged 20-75 years at enrollment
3. History of edentulism in the study area of at least two months
4. Neighboring tooth/teeth to the planned crown(s) must have natural root(s)
5. Presence of natural teeth, partial prosthesis and/or implants in the opposite jaw in contact with the planned crowns
6. Deemed by the investigator to have a bone height and width suitable for 3.0 mm diameter study implant
7. Deemed by the investigator as likely to present an initially stable implant situation

Exclusion Criteria:

1. Unlikely to be able to comply with study procedures, as judged by the investigator
2. Uncontrolled pathologic processes in the oral cavity
3. Known or suspected current malignancy
4. History of radiation therapy in the head and neck region
5. History of chemotherapy within 5 years prior to surgery
6. Systemic or local disease or condition that could compromise post-operative healing and/or osseointegration, as deemed by the investigator
7. Uncontrolled diabetes mellitus
8. Corticosteroids or any other medication that could influence post-operative healing and/or osseointegration
9. Smoking more than 10 cigarettes per day
10. Present alcohol and/or drug abuse
11. Involvement in the planning and conduct of the study (applies to both Astra Tech staff and staff at the study site)
12. Previous enrollment in the present study
13. Simultaneous participation in another clinical study, or participation in a clinical study during the last weeks prior to enrollment

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2011-06 (Actual); Primary Completion 2014-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Li Dehua, Prof, Principal Investigator — Dept. of Oral Implants, School of Stomatology, Fourth Military Medical University, Xi'an
Locations (3):
- China (3):
  - Tong Ji University, Oral Implants Department, Shanghai
  - School of Stomatology Wuhan University, Wuhan
  - Dept. of Oral Implants, School of Stomatology, Fourth Military Medical University, Xi'an

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Implants
Period: Overall Study
Arm/Group | OsseoSpeed™ TX
Started | 45; 47 Implants
Completed | 40; 42 Implants
Not Completed | 5; 5 Implants
Not completed — Lost to Follow-up | 5

BASELINE CHARACTERISTICS:
Arm/Group | OsseoSpeed™ TX
Number analyzed (Participants) | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.4 (14.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 21
Region of Enrollment [Number; unit: participants]
  China | 45

OUTCOME MEASURES:

1. Primary Outcome: Implant Survival
Description: Implant survival rate evaluated clinically and radiographically.
Time Frame: Measured at the 3-year follow-up visit after implant loading.
Population: Intention to treat (ITT), including all participants that received at least one implant, a total of 45 subjects (47 implants).
  A total of 5 subjects (5 implants) had been lost to follow-up at time of the 3-year follow-up visit, giving an overall number of 40 subjects (42 implants) as basis for the analysis of three year survival rate.
Measure: Count of Units; unit: Implants
Units Other Than Participants: Implants
Arm/Group | OsseoSpeed™ TX
Number analyzed (Participants) | 40
Number analyzed (Implants) | 42
Implants | 42

2. Secondary Outcome: Implant Stability
Description: Implant stability evaluated clinically/manually (recorded as stable yes/no).
Time Frame: Measured at the 3-year follow-up visit after implant loading.
Population: 40 subjects (42 implants) completed the 3-year follow-up visit. Analysis of implant stability was performed on the All Patients Treated (APT) population.
Measure: Count of Units; unit: implants
Units Other Than Participants: implants
Arm/Group | OsseoSpeed™ TX
Number analyzed (Participants) | 40
Number analyzed (implants) | 42
implants | 42

3. Secondary Outcome: Marginal Bone Level Alteration
Description: Marginal Bone Level (mm) determined from radiographs and expressed as a difference from a reference point on the implant to the most coronal bone-to-implant contact on the mesial and distal aspect of the implant.
  Marginal Bone Level expressed in millimeters obtained at the 3-year follow-up visit compared to values obtained at delivery of the temporary restoration i.e. loading (baseline).
Time Frame: Measured at the 3-year follow-up visit after implant loading.
Population: 40 subjects (42 implants) completed the 3-year follow-up visit. Protocol deviations were excluded (9 subjects, 10 implants), giving a per-protocol analysis population of 31 subjects (32 implants).
Measure: Mean (Standard Deviation); unit: millimeter
Units Other Than Participants: Implants
Arm/Group | OsseoSpeed™ TX
Number analyzed (Participants) | 31
Number analyzed (Implants) | 32
millimeter | 0.52 (0.84)

4. Secondary Outcome: Condition of the Periimplant Mucosa by Assessment of Probing Pocket Depth (PPD).
Description: Change in pocket depth expressed in millimeters at time of the 3 years follow-up visit, compared to values obtained at delivery of permanent restoration, i.e. loading (baseline).
  Negative value = increased pocket depth.
Time Frame: Measured at implant loading and at the 3-year follow-up visit after loading.
Population: 40 subjects (42 implants) completed the 3 years follow-up visit. Protocol deviations were excluded (9 subjects, 10 implants), giving a per-protocol analysis population of 31 subjects (32 implants).
Measure: Mean (Standard Deviation); unit: millimeter
Units Other Than Participants: Implants
Arm/Group | OsseoSpeed™ TX
Number analyzed (Participants) | 31
Number analyzed (Implants) | 32
millimeter | -0.26 (0.73)

5. Secondary Outcome: Condition of the Periimplant Mucosa by Assessment of Bleeding on Probing (BoP).
Description: Condition of the periimplant mucosa by assessment of Bleeding on Probing (BoP). Presented as % of implants that show presence of bleeding on probing at time of the 3-year follow-up visit.
Time Frame: Measured at implant loading and at the 3-year follow-up visit after loading.
Population: as for outcome 3
Measure: Count of Units; unit: implants
Units Other Than Participants: implants
Arm/Group | OsseoSpeed™ TX
Number analyzed (Participants) | 31
Number analyzed (implants) | 32
implants | 2

6. Secondary Outcome: Presence of Plaque
Description: Occurence of plaque around the study implant. Presented as proportion of implants that show presence of plaque at time of the 3-year follow-up visit.
Time Frame: Measured at the 3-year follow-up visit after implant loading.
Population: as for outcome 3
Measure: Count of Units; unit: implants
Units Other Than Participants: implants
Arm/Group | OsseoSpeed™ TX
Number analyzed (Participants) | 31
Number analyzed (implants) | 32
implants | 2

7. Secondary Outcome: Gingival Zenith Score
Description: Gingival zenith score measured from the gingival zenith to the incisal edge of the prosthetic crown with a periodontal probe to nearest 0.5 mm.
  Presented as change from loading of permanent restoration to time of the 3-year follow-up visit.
Time Frame: Measured at implant loading and at the 3-year follow-up visit after loading.
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: millimeter
Units Other Than Participants: implants
Arm/Group | OsseoSpeed™ TX
Number analyzed (Participants) | 31
Number analyzed (implants) | 32
millimeter | -0.03 (0.74)

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | OsseoSpeed™ TX
Serious Adverse Events (participants affected / at risk) | 0/45
Other Adverse Events (participants affected / at risk) | 0/45

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less